CLINICAL TRIAL: NCT05975710
Title: Textbook and Survival Outcomes of Minimally Invasive Pancreatoduodenectomy : A Retrospective Multicenter Analysis of 1,552 Patients in Korean Study Group on Minimally Invasive Pancreatic Surgery (K-MIPS)
Brief Title: Textbook and Survival Outcomes of MIPD in South Korea
Status: Completed | Type: Observational
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Song Cheol Kim, Professor, Asan Medical Center
Other Study IDs: KMIPS
Record Dates: First submitted 2023-07-15; First posted 2023-08-04 (Actual); Last update posted 2023-08-04 (Actual); Status verified 2023-08

CONDITIONS: Surgery-Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this study was to investigate the current status of minimally invasive pancreatoduodenectomy (MIPD) in South Korea with regard to demographics, perioperative outcomes, risk factors for textbook outcome of pancreatic surgery (TOPS) and survival outcomes of periampullary cancer.

DETAILED DESCRIPTION:
Pancreatoduodenectomy (PD) is the most complicated abdominal surgical procedure and in addition, the difficulty of this operation is much higher if it is performed using minimally invasive methods. Since these first minimally invasive pancreatoduodenectomy (MIPD) surgeries were performed, they have been adopted by various institutions and their effectiveness has been highlighted in several studies. Advantages of MIPD include a short hospital stay, less blood loss, and less pain compared to open procedures. However, a multicenter randomized controlled trial that compared LPD and open pancreatoduodenectomy (OPD) reported that LPD had a higher complication-related mortality rate than OPD. Meta-analysis of randomized controlled trials of LPD versus OPD also reported that LPD had no advantage over OPD but with a high risk of bias and moderate to low level of evidence. In a meta-analysis of RPD and OPD, RPD was found to have the advantages of less blood loss, shorter hospital stay, and lower wound infection rate than OPD, but to date, no studies have reported results for randomized controlled trials of RPD. Although it is still early to make generalized conclusions about MIPD due to the selection bias inherent in retrospective studies and an insufficient number of prospective studies, the frequency with which MIPD is being performed is gradually increasing. Studies on the learning curve of MIPD are currently in progress, and one study recommended establishment of an MIPD registry for research purposes. South Korea is one of the country leading the implementation of MIPD, and several Korean groups have published studies on this surgery and have collaborated to establish a registry in line with global trends. After the establishment of the Korean study group on Minimally Invasive Pancreatic Surgery (K-MIPS) in 2019 (http://kmips.or.kr/index.html), 1,552 MIPD patients were retrospectively enrolled. Apart from this, the textbook outcomes after surgery was recently emerged as a valuable approach for assessing surgical success, as it considers multiple quality measures to provide a comprehensive indication of overall outcomes. Recently, the Dutch Pancreatic Cancer Group reported about textbook outcome of pancreatic surgery (TOPS), which is also a multidimensional measure that allows assessment of the quality of surgical outcomes, and several papers have investigated textbook outcome after hepatobiliary and pancreatic surgery. From this perspective, conducting an analysis of the current status of MIPD in Korea and evaluating the surgical outcomes by TOPS would provide valuable insights, making this study highly relevant and meaningful. The aim of this study was to describe the current status of MIPD in South Korea in terms of demographics, perioperative outcomes, survival outcomes, TOPS and risk factor of TOPS. In addition, current study compared subgroups classified according to hospital volume in South Korea to determine if hospital volume affects perioperative outcomes.

ELIGIBILITY:
Inclusion Criteria:

The patients who underwent MIPD between May 2007 and April 2020 at ten tertiary referral institutions in South Korea.

Exclusion Criteria:

None

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: This retrospective multicenter cohort study evaluated 1,552 patients who underwent MIPD by 24 experienced pancreatic surgeons between May 2007 and April 2020 at ten tertiary referral institutions in South Korea. The research was conducted using data registered in the registry of the Korean study group on Minimally Invasive Pancreatic Surgery (K-MIPS). The consecutive patient's data were recorded retrospectively and self-registered at each institution.
Sampling Method: Non-Probability Sample
Enrollment: 1552 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Success rate of textbook outcome of pancreatic surgery | 3 months
  If none of the seven specified factors (1. postoperative pancreatic fistula, 2. bile leakage, 3. postpancreatectomy hemorrhage, 4. Clavien-Dindo 3 or higher of complications, 5. readmission within 90 days, 6. in-hospital or 90-day mortality, 7. postoperative hospital stay of more than 14 days) occur after minimally invasive pancreatoduodenectomy, it is defined as TOPS success in current study.
  In other words, a patient's outcome is considered successful if they do not experience any of these adverse events or complications within the specified time frames.

CONTACTS AND LOCATIONS:
Overall Officials: Song Cheol Kim, MD.PhD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan medical center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No